CLINICAL TRIAL: NCT02417363
Title: Affiliated Hospital of Stomatology, School of Medicine, Zhejiang University
Brief Title: Study on the Relationship Between Periodontitis and Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Na Zhou, The stomatological hospital affiliated to medical college, Zhejiang University, Zhejiang University
Other Study IDs: ZJUSH2015-1
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Periodontitis
Keywords: biomarkers; renal disease; periodontitis
MeSH Terms: conditions — Periodontitis; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples are placed into 1.5 ml Eppendorf tubes and maintained at -70℃ for further analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group A: the control group,healthy individuals
- Group B: patients with 1-4 stage K/DOQI (Kidney Disease Outcome Quality Initiative) chronic kidney disease, but healthy periodontium
- Group C: patients with periodontitis, but healthy renal conditions
- Group D: patients with 1-4 stage K/DOQI (Kidney Disease Outcome Quality Initiative) chronic kidney disease and periodontitis

SUMMARY:
Analysis of inflammatory markers in periodontitis and patients with early and middle stage renal disease.

DETAILED DESCRIPTION:
A total of 200 population is recruited, individuals are divided into four groups according to a periodontal examination and a general physical examination: healthy individuals ,periodontitis, renal disease patients with healthy periodontium, and renal disease patients wth peridontitis. Fasting blood samples and gingival crevicular fluid are collected from all individuals, and inflammatory markers are analysed for the four groups.

ELIGIBILITY:
Inclusion Criteria:

* all participants were in general good health(except renal disease) and non-smoking

Exclusion Criteria:

* less than 20 teeth in the dentin
* hypertension
* the presence of systemic disease (e.g., diabetes mellitus ,coronary heart disease, liver, or lung disease)
* a history or the symptom of any other acute or chronic infections
* systemic antibiotic treatment within previous 4 weeks
* periodontal treatment within1 month

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 individuals are recruited for each group, the factors of age and gender are matched while selecting the incruited indiduals,all participants were in general good health(except renal disease) and non-smoking.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers analysis of the four groups | 3 months after sampling
  Analysis of inflammatory biomarkers of blood and gingival crevicular fluid samples of the four groups

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, Study Director — Affiliated Hospital of Stomatology, School of Medicine, Zhejiang University
Locations (1):
- Affiliated Hospital of Stomatology, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China